CLINICAL TRIAL: NCT02173808
Title: A Phase I Study to Evaluate the Pharmacokinetic and Pharmacodynamic Profile of a Single Injection of Levonorgestrel Butanoate (LB) for Female Contraception
Brief Title: A Phase I Study to Evaluate the PK and PD of a Single Injection of Levonorgestrel Butanoate for Female Contraception
Acronym: CCN011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCN011
Record Dates: First submitted 2014-05-12; First posted 2014-06-25 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2014-04

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior | interventions — levonorgestrel butanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contraceptive (Experimental)
  Interventions: Biological: levonorgestrel butanoate

INTERVENTIONS:
Biological: levonorgestrel butanoate

SUMMARY:
To evaluate the levonorgestrel (LNG) pharmacokinetic (PK) profile following injection of a single 20 mg dose of levonorgestrel butanoate (LB).

DETAILED DESCRIPTION:
This is a Phase I single center, open-label, single dose pharmacokinetic and pharmacodynamic study of an injectable formulation of levonorgestrel butanoate (LB) jointly developed by the National Institute of Child Health and Human Development (NICHD) and CONRAD, and manufactured by Coldstream Laboratories, Inc. Healthy normal weight and obese women will be followed as outpatients for up to eight months. During this study, subjects will undergo a screening cycle to confirm normal ovulatory function, and then receive active treatment with a single injection of LB. They will undergo frequent evaluations to obtain serum samples to evaluate drug levels and ovulatory function, as well as transvaginal ultrasound and cervical mucus evaluation at selected visits. Follow up will continue until normal ovulatory cycles resume. Based upon detailed studies in non-human primates, it is expected that most subjects will resume menstrual cyclicity within 12- 26 weeks following the injection. Subjects will continue to be followed for one normal cycle after return of menses. This study will be conducted by the NICHD at one of the Contraceptive Clinical Trials Network (CCTN) sites (Oregon Health & Science University, (OHSU)) in the USA and will enroll approximately 16 women.

This study will enroll approximately 16 subjects that demonstrate favorable cervical mucus and normal ovulatory function during a baseline cycle. Enrollment will be stratified to ensure that 50% of the subjects have a BMI >32 kg/m2 and <40 kg/m2 and approximately 50% of subjects have a BMI <32 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health
2. Aged 18-44 years, inclusive, at the enrollment visit
3. Intact uterus with at least one ovary
4. Serum progesterone value ≥ 3 ng/mL at the Screening Visit (V0-P)
5. Pap test within the last 12 months or undergo a Pap test at screening prior to enrollment. If a potential subject states that she has had a Pap test within the last 12 months, then she will need to provide documentation of acceptable test results
6. Cervical mucus score of >7, which is based on the modified Insler scoring system during the screening cycle. The cervical mucus is collected by aspiration and the assessment is based on the modified Insler scoring system (the volume and pH of the mucus are not included in the total scoring) yielding a total possible score of 12 (3, 4)
7. Regular menstrual cycles that occur every 24 - 35 days

   1. If subject is postpartum or post-abortal (with abortion in second trimester), she will be required to have two normal menstrual cycles prior to screening
   2. If subject had an abortion in the first trimester, she will be required to have at least one menstrual cycle (two menses) prior to screening
8. Heterosexually abstinent or, if heterosexually active, must have undergone previous tubal sterilization, be in monogamous relationship with a vasectomized partner, or only use male or female condoms (use of condoms that are pre-lubricated with or without spermicide is acceptable) for the entire duration of the study. Use of a spermicide applied separately is not allowed. Cervical caps or diaphragms are not allowed during study participation
9. In the opinion of the investigator, able to comply with the protocol, willing to record requested information in the daily diary, and live within the study site catchment area or within a reasonable distance from the site
10. Understand and sign an IRB approved informed consent form prior to screening activities (including fasting blood draw)
11. Willing to refrain from use of any vaginal creams, lubricants, gels, or spermicides for 3 days prior to study admission through to the end of the study
12. Agree not to participate in any other clinical trials during the course of this study

Exclusion Criteria:

1. Known hypersensitivity or contraindication to progestins
2. Known or suspected pregnancy
3. Prior hysterectomy or bilateral oophorectomy
4. Prior cervical surgery (LEEP, Cone biopsy)
5. A history (within prior 12 months) of drug or alcohol abuse
6. Undiagnosed abnormal genital bleeding
7. Undiagnosed vaginal discharge or vaginal lesions or abnormalities. Subjects diagnosed at screening with a Chlamydia or gonococcus infection may not be included in the trial unless they are treated and proof of cure is documented after treatment (i.e. repeat test with negative results). In accordance with PI/medical designee assessment and local standards of practice, women with a history of genital herpes can be included if outbreaks are infrequent. Antiviral prophylactic therapy is permitted
8. Uncontrolled thyroid disorder
9. Any Pap test finding that would require additional workup or treatment during the study interval. HPV testing will not be done at screening for these subjects
10. Use of an injectable hormonal contraceptive (Depo-Provera®) within the past 10 months
11. Use of oral contraceptives, contraceptive implants, or other sex steroid hormones within 30 days prior to screening visit
12. Women who are breastfeeding or within 30 days of discontinuing breast feeding
13. Women planning to undergo major surgery within four months of study enrollment
14. Women planning pregnancy within their months of study enrollment
15. Smoking in women who are ages 18-44 years old that smoke 15 cigarettes or more per day must be evaluated by the PI for inclusion based on risk factors that would increase their risk for cardiovascular (CVD) and thromboembolism
16. Current or past deep vein thrombophlebitis or thromboembolic disorders
17. History of known thrombophilia in a first-degree relative <45 years of age suggesting familial defect in blood coagulation system, which in the opinion of the principal investigator, suggests use of a hormonal contraceptive could pose a significant risk
18. Cerebrovascular or cardiovascular disease or increased risk for arterial thrombosis
19. History of retinal vascular lesions, unexplained partial or complete loss of vision
20. Known or suspected carcinoma of the breast, endometrium, or any other known or suspected progestin-dependent neoplasia
21. Past history of any other carcinoma (excluding basal cell carcinomas) unless in remission for more than 5 years
22. Current or past medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by use of a hormonal contraceptive, unless she is stable on antidepressant medication
23. Headaches with focal neurological symptoms only in women over 35 years old
24. History of cholestatic jaundice of pregnancy or jaundice with prior steroid use or other benign or malignant liver tumors; active liver disease
25. Systolic BP > 140 mm Hg and/or Diastolic blood pressure (BP) > 90 mm Hg after 5-10 minutes rest
26. Clinically significant abnormal serum chemistry values according to the Principal Investigator's judgment
27. Participation in another clinical trial involving an investigational drug or device within last 30 days (prior to screening)
28. Use of liver enzyme inducers within last 90 days (prior to screening) or intention to use liver enzyme inducers during the study
29. Known HIV infection
30. Women at high risk of contracting HIV, e.g. women with multiple sex partners who need to use condoms consistently, injection drug users. Women enrolled in the study, who use condoms to protect against STIs or pregnancy, should be instructed that they can use condoms that are pre-lubricated with spermicide or lubricated, but they cannot use a spermicide applied separately and they should record all condom use in their diaries
31. Women who use any medications on the Exclusionary Medication List OR used any within the past three months prior to the screening visit
32. Women with BMI ≥40 kg/m2 are excluded
33. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PK profile will be assessed in terms of the pharmacodynamics profile that correlates with the goal of reversible female contraception. | May 2011 - June 2012 (13 months)
  PK profile will be assessed in terms of the pharmacodynamics profile that correlates with the goal of reversible female contraception. For each subject and for the low and high BMI groups, the primary endpoint will be the time to return of ovulation based on two consecutive serum progesterone >3 ng/L or a single progesterone >10 ng/L.

SECONDARY OUTCOMES:
Assessing the pharmacodynamics (PD) profile through evaluation of endometrial thickness, ovarian follicular development, cervical mucus changes, steroid hormones, gonadotropins and sex hormone binding globulin. | May 2011 - June 2012 (13 months)
Assessing the pharmacodynamics (PD) profile through evaluation of ovarian follicular development. | May 2011 - June 2012 (13 months)
Assessing the pharmacodynamics (PD) profile through evaluation of cervical mucus changes. | May 2011 - June 2012 (13 months)
Assessing the pharmacodynamics (PD) profile through evaluation of steroid hormones. | May 2011 - June 2012 (13 months)
Assessing the pharmacodynamics (PD) profile through evaluation of gonadotropins. | May 2011 - June 2012 (13 months)
Assessing the pharmacodynamics (PD) profile through evaluation of sex hormone binding globulin. | May 2011 - June 2012 (13 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States